CLINICAL TRIAL: NCT03785899
Title: Automatic Oxygen Control (SPOC) in Preterm Infants - Evaluation of a Revised Algorithm and Effect of Averaging Time of Pulse Oximetry Signal
Brief Title: Automatic Oxygen Control (SPOC) in Preterm Infants
Acronym: optimalSPOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Fritz Stephan GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: optimalSPOC
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-08

CONDITIONS: Infantile Respiratory Distress Syndrome; Ventilator Lung; Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RMC only (No Intervention): routine manual control (RMC) of the fraction of inspired oxygen (FIO2)
- SPOCnew and 2s SpO2 averaging (Experimental): routine manual control (RMC) + automatic oxygen control (SPOC) with "new" algorithm of the fraction of inspired oxygen (FIO2).
  The SpO2 signal averaging time is 2s.
  Interventions: Device: SPOCnew; Device: 2s SpO2 averaging
- SPOCnew and 8s SpO2 averaging (Experimental): routine manual control (RMC) + automatic oxygen control (SPOC) with "new" algorithm of the fraction of inspired oxygen (FIO2).
  The SpO2 signal averaging time is 8s.
  Interventions: Device: SPOCnew; Device: 8s SpO2 averaging
- SPOCold and 2s SpO2 averaging (Active Comparator): routine manual control (RMC) + automatic oxygen control (SPOC) with "old" algorithm of the fraction of inspired oxygen (FIO2).
  The SpO2 signal averaging time is 2s.
  Interventions: Device: SPOCold; Device: 2s SpO2 averaging
- SPOCold and 8s SpO2 averaging (Active Comparator): routine manual control (RMC) + automatic oxygen control (SPOC) with "old" algorithm of the fraction of inspired oxygen (FIO2).
  The SpO2 signal averaging time is 8s.
  Interventions: Device: 8s SpO2 averaging; Device: SPOCold

INTERVENTIONS:
Device: SPOCnew — SPOC is an automated, algorithm based adjustment of the fraction of inspired oxygen in relation to arterial saturation (SPO2). The revised "new" algorithm is turned on.
  Arms: SPOCnew and 2s SpO2 averaging; SPOCnew and 8s SpO2 averaging
Device: 8s SpO2 averaging — The arterial saturation (SPO2) will be averaged over 8s.
  Arms: SPOCnew and 8s SpO2 averaging; SPOCold and 8s SpO2 averaging
Device: SPOCold — SPOC is an automated, algorithm based adjustment of the fraction of inspired oxygen in relation to arterial saturation (SPO2). The former "old" algorithm is turned on.
  Arms: SPOCold and 2s SpO2 averaging; SPOCold and 8s SpO2 averaging
Device: 2s SpO2 averaging — The arterial saturation (SPO2) will be averaged over 2s.
  Arms: SPOCnew and 2s SpO2 averaging; SPOCold and 2s SpO2 averaging

SUMMARY:
Single-center, randomised controlled, cross-over clinical trial in preterm infants born at gestational age below 34+1/7 weeks receiving supplemental oxygen and respiratory support (continous positive airway pressure (CPAP) or non-invasive ventilation (NIV) or invasive ventilation (IV)). Routine manual control (RMC) of the fraction of inspired oxygen (FiO2) will be tested against RMC supported by automatic control (SPOC) with "old"-algorithm and RMC supported by CLAC with "new"-algorithm.

The first primary hypothesis is, that the use of the "new" algorithm results in more time within arterial oxygen saturation (SpO2) target range compared to RMC only. The a-priori subordinate hypothesis is, that the new algorithm results in more time within SpO2 target range compared to SPOCold.

The second primary hypothesis is, that the use of 2 seconds averaging time of the SpO2 Signal results in more time within arterial oxygen saturation (SpO2) target range compared to the use of 8 seconds averaging interval of the SpO2 signal.

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVE In preterm infants receiving supplemental oxygen, routine manual control (RMC) of the fraction of inspired oxygen (FiO2) is often difficult and time consuming. The investigators developed a system for closed-loop automatic control (SPOC) of the FiO2. The objective of this study is to test a revised, "new" algorithm with 3 adaptions against the former "old" algorithm and against RMC. The 3 adaptions are:

1. Faster re-adjustment to baseline-FiO2 (baseline FiO2: mean FiO2 during the previous 5min)
2. Delayed reduction of FiO2 below baseline FiO2
3. Maximum FiO2 adjustable by user

The first primary hypothesis is, that the application of SPOCnew in addition to RMC results in more time within arterial oxygen saturation (SpO2) target range compared to RMC only. The a-priori subordinate hypothesis is, that the revised algorithm is more effective as the old algorithm to maintain the SpO2 in the target range.

The second primary hypothesis is, that the shortening of averaging time used for the SpO2 Signal from 8 seconds to 2 seconds results in more time within SpO2 target range for both, SPOCnew and SPOCold.

Further hypotheses for exploratory testing are, that the SPOC new algorithm will achieve a lower proportion of time with SpO2 above and below the target range, hyper- and hypoxia and an improved stability of cerebral oxygenation (measured as rcStO2 and rcFtO2E determined by Near-infrared spectroscopy) compared with SPOCold and RMC. Reduction of staff workload (estimated by number of manual adjustments per hour) by SPOC. Validation of a clinical scoring tool to monitor severity of apnea of prematurity.

STUDY DESIGN The Study is designed as a single-center, randomized controlled, cross-over clinical trial in preterm infants receiving mechanical ventilation or nasal continuous positive airway pressure or non-invasive ventilation and supplemental oxygen (FiO2 above 0.21). Within a 30-hour period the investigators will compare 6 hours of RMC with 12-hour periods of RMC supported by SPOCnew algorithm or SPOCold algorithm, respectively. During intervals with SPOC control the SpO2 Signal averaging time will be 2 second or 8seconds , respectively, for 6 hours each.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth <34+1/7weeks and
* invasive mechanical ventilation OR noninvasive ventilation OR continous positive airway pressure support and
* Fraction of inspired oxygen above 0.21 before inclusion and
* more than 2 hypoxaemic events (arterial oxygen saturation below 80%) within 8 hours before inclusion and
* parental written informed consent

Exclusion Criteria (any of the following):

* congenital pulmonary anomalies
* congenital heart defects influencing SpO2 (i.e. cyanotic heart defects)
* right-to -left shunt through a PDA
* Severe neonatal complications during study period (sepsis, necrotising enterocolitis)
* diaphragmatic hernia or other diaphragmatic disorders

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of time with SpO2 within target range | 30 hours
  Comparison of proportion of time with SpO2 within target range and time above target range if no supplemental oxygen was administered at that time and within the preceding 30sec between the five treatment modalities

SECONDARY OUTCOMES:
Proportion of Time with SpO2 above target range | 30 hours
  Comparison of proportion of time with SpO2 above target range if supplemental oxygen was administered at that time or within the preceding 30sec .
Proportion of Time with SpO2 below target range | 30 hours
  Comparison of proportion of time with SpO2 below target range.
Proportion of Time with Hypoxia | 30 hours
  Comparison of proportion of time with SpO2 below 80%.
Proportion of Time with Hyperoxia | 30 hours
  Comparison of proportion of time with SpO2 above 97% if supplemental oxygen was administered at that time or at anytime during the previous 30 seconds.
Stability of cerebral oxygenation | 30 hours
  "Area under the curve" of cerebral tissue saturation or fraction of tissue oxygen extraction outside of the infants Median +- 5% or outside of the "safe" interval of 55-80% rcStO2.
Severe hypoxemic episodes | 30 hours
  Rate of episodes with SpO2 <80% for at least 60seconds

OTHER OUTCOMES:
Staff workload | 30 hours
  number of manual adjustments of inspired oxygen per time
Validation of clinical Apnea Score | 30 hours
  Validation of a modified Apnea Score monitored by clinical staff by correlation between Score and other secondary outcomes. The modified Apnoea Score aims to quantify the burden from apnoea-bradycardia-syndrome by assigning 1-2-4 or 8 points according to event severity. Points are summed up during each treatment period in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph E Schwarz, MD, Principal Investigator — University of Tubingen, University Hospital, Dept. Neonatology
Locations (1):
- Department of Neonatology, University Children's Hospital, Tübingen, Germany

REFERENCES:
- [Derived] Langanky LO, Kreutzer KB, Poets CF, Franz AR, Schwarz CE. Pulse oximetry signal loss during hypoxic episodes in preterm infants receiving automated oxygen control. Eur J Pediatr. 2024 Jul;183(7):2865-2869. doi: 10.1007/s00431-024-05549-9. Epub 2024 Apr 9. PMID 38592485
- [Derived] Schwarz CE, Kreutzer KB, Langanky L, Wolf NS, Braun W, O'Sullivan MP, Poets CF, Franz AR. Randomised crossover trial comparing algorithms and averaging times for automatic oxygen control in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2022 Jul;107(4):425-430. doi: 10.1136/archdischild-2021-322096. Epub 2021 Nov 24. PMID 34819347